CLINICAL TRIAL: NCT06764043
Title: Molar-Incisor Hypomineralization (MIH) Vs Periodontal Health: Evaluation of Clinical Periodontal Indexes and Biomarkers (MMP-8, MMP-20 and TGF- Β1)
Brief Title: Molar-Incisor Hypomineralization Vs Periodontal Health
Acronym: MIH
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, DİLARA NİL GÜNAÇAR, Assoc.Prof., Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2023/121; 1495 (Other Grant/Funding Number: Recep Tayyip Erdogan University, Department of Scientific Research Project)
Record Dates: First submitted 2024-12-24; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Molar-Incisor Hypomineralization; Peridontal Disease
Keywords: Gingival crevicular fluid; Matrix metalloproteinase 8; Matrix metalloproteinase 20
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Clinical evaluation — In this study, it was aimed to measure the levels of MMP-8, MMP-20, and TGF-β1 in GCF together with the volume of GCF to investigate the effect of MIH on oral hygiene, and gingival health, and also to evaluate the relationship between MIH, and various biomarkers.

SUMMARY:
Background: To investigate the effect of molar incisor hypomineralization (MIH) on periodontal health, to evaluate the relationship between gingival crevicular fluid (GCF) volume, and GCF biomarkers such as matrix metalloproteinase-8 (MMP-8), matrix metalloproteinase-20 (MMP-20), and transforming growth factor-beta 1 (TGF-β1), and MIH.

Methods: The study was conducted on 40 pediatric patients diagnosed with MIH (Study Group/SG), and 40 pediatric patients healthy for MIH (Control Group/CG). Clinical periodontal measurements (plaque index (PI), gingival index (GI), probing pocket depth (PPD), and GCF volume were performed. Concentrations of MMP-8, MMP-20, and TGF-β1 in GCF were determined using enzyme-linked immunosorbent assay (ELISA). Mann-Whitney U test and T-test were used for comparisons between groups. Significance was set at p=0.05 for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* the ages of 8 and 14 who were diagnosed with MIH in their maxillary permanent first molars,
* had healthy maxillary permanent first molars,
* scored 3 (positive) or 4 (definitely positive) on the Frankl Behavior Scale,
* had no mental or physical disability,
* did not need urgent treatment and/or were not in pain,
* agreed to participate in the study with their parents and signed the consent form.

Exclusion Criteria:

* Children with systemic, chronic, and/ or metabolic diseases,
* under active orthodontic treatment, with developmental defects of enamel (excluding MIH), or born prematurely

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric population with MIH
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Periodontal indexes measurement | 1 day
  PI, GI, and PPD measurements were performed to evaluate the periodontal health of the children participating in the study.
GCF measurement | 1 day
  In the study, GCF was collected in the morning hours (between 09:00 and 11:00) one day after the patient's clinical periodontal measurements were complete.
Evaluation of MMP-8, MMP-20 and TGF-β1 Levels by ELISA Method | for three days from the beginning of the study
  The levels of MMP-8 (Elabscience® EL-H1450, Biotechnology Co., Ltd, Wuhan, China), MMP-20 (Bioassay Technology Laboratory, Cat. No E4139Hu), and TGF-β1 (Elabscience® EL-H0110, Biotechnology Co., Ltd, Wuhan, China) in GCF samples were measured using ELISA kits.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdoğan University Faculty of Dentistry, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bilgir BS, Aydinoglu S, Arslan I, Atak M, Kose O, Gunacar DN. Analysis of MMP-8, MMP-20, and TGF-beta1 in molar-incisor hypomineralization and assessment of periodontal health. BMC Oral Health. 2025 Jul 17;25(1):1189. doi: 10.1186/s12903-025-06551-9. PMID 40676550